CLINICAL TRIAL: NCT03390868
Title: Effects of a Web-based Training Programme for Professional Carers Working With People With Learning Disabilities Who Exhibit Challenging Behaviour
Brief Title: Effects of a Web-based Training Programme Focusing on Challenging Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University West, Sweden (Other)
Responsible Party: Principal Investigator, Helena Antonsson, Senior lecturer, med dr., Umeå University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Challenging behaviour
Record Dates: First submitted 2017-12-29; First posted 2018-01-04 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Challenging Behaviour
Keywords: Interaction; challenging behaviour; training

STUDY DESIGN:
Intervention Model Description: Intervention arm: web-based training for staff working with people with intellectuall disabilities and challenging behaviour Other: control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Phase 1, participants in the intervention group will take part in an web-based training for staff working with people with intellectual disabilities and challenging behaviour aiming to in a more effective way communicate to prevent challenging behaviour. The participants (staff) will by their own, go through the web-based training program during working hours. Measurement are conducted before intervention, at intervention completion an average of 12 weeks, and for a 3 month follow up after completed intervention
  Interventions: Behavioral: Web-based training for staff
- control arm (Other): Control arm: participants in the control-group will maintain regular care and have the opportunity to receive the web-based training for staff working with people with intellectual disabilities and challenging behaviour in phase 2.
  Interventions: Behavioral: Web-based training for staff

INTERVENTIONS:
Behavioral: Web-based training for staff — This web-based training program is focusing on strengthening the carers' communication skills. Video lectures on the definitions, characteristics and causes of challenging behavior will be given. Video lectures will also be given on the importance of the carers' views on their values, emotions, abilities and attitude towards people with intellectual disabilities and on the impact that workplace culture and environmental factors have on the quality of interactions. The program also includes written cases that gives the participants opportunities to reflect upon approaches supporting a successful interaction. It also covers factors to consider when mental illness and challenging behavior occur. The time to complete the web-based training program is estimated at approximately ten hours.

SUMMARY:
The interaction between people with intellectual disabilities and professional carers is often influenced by communicative difficulties contributing challenging behaviours.

Aim: The aim of this study is to evaluate a web-based training program aimed at improving carers' abilities to interact with people with learning disabilities who exhibit challenging behaviours and to explore carers' experiences of participating in such a program.

Method: This study has a cross-sectional design. Sample: The study will be conducted in twenty special community-based accommodations, group-homes, in Sweden that each houses 4-8 residents. The staff in the group-homes is working independently with the manager located at distance.The staff (N=221) in this study works with people with intellectual disabilities who has different functional levels, from moderate to profound intellectual disabilities. They have different educational backgrounds: from basic nursing education at the college level to university degree.

Intervention: The intervention consists of a web-based training program, available for all staff working in special accommodations for people with intellectual disabilities. The web-based training program focuses on strengthening the carers' communication skills.

Procedure: The social Services authorities and the managers from each home agreed to the project. The carers have given their informed consent to attend the study. The participants will by their own during working hour go through the web-based program. The time to complete the web-based training program is estimated at approximately ten hours.

Data-analysis: Descriptive statistics will be used for demographic data. Proportions will be compared to the chi-square test. The mean values between the groups will be compared by t-test or Mann-Whitney's U-test, as appropriate. Changes in the mean between and in the groups will be compared with paired t-test. Double-sided significance test will be used throughout. Data will be presented at a group level.

DETAILED DESCRIPTION:
A literature review shows that the interaction between adult persons with intellectual disabilities and professional carers is a complex combination of verbal and non-verbal expressions. Attempts to communicate often lead to misunderstandings from both parties, as well as challenging behaviors such as aggression and violence. The literature shows that challenging behavior often leads to physical constraints. Literature studies also emphasize the importance of education, knowledge and support for staff. Therefore, we want to investigate whether it is possible to reduce challenging behavior through education on causes of challenging behavior and successful interaction for carers in special housing.

Aim: To study the effects of a web-based training program to increase staff's ability to better communicate and interact with persons with intellectual disabilities and challenging behaviors.

Method: The study has a cross-sectional design.

Intervention: The intervention was inspired by an evidence-based conceptual model for staff training in challenging behaviour. The intervention consists of a web-based training program, available for all carers working in special accommodations for people with intellectual disabilities.

The web-based training program focuses on strengthening the carers' communication skills. Video lectures on the definitions, characteristics and causes of challenging behaviour will be given. Video lectures will also be given on the importance of the carers' views on their values, emotions, abilities and attitude towards people with intellectual disabilities, and on the impact that workplace culture and environmental factors have on the quality of interactions. The web-based training program also includes written cases that gives the participants an opportunity to reflect upon approaches supporting a successful interaction. It also covers factors to consider when mental illness and challenging behaviour occur. The web-based training program includes the opportunity to follow the carers' activity regarding time and frequency of studying. The time to complete the web-based training program is estimated at approximately ten hours.

Context: The study will be conducted in twenty special community-based accommodations, group-homes, in Sweden that each houses 4-8 residents. The residents has their own private rooms, but shares a communal space with a living room and a kitchen with a dining table. The staff in the group-homes is working independently with the manager located at distance.

Participants:The carers in this study works with people with intellectual disabilities who has different functional levels, from moderate to profound intellectual disabilities. They have different educational backgrounds: from basic nursing education at the college level to university degree.

Procedure: Prior to handing out the questionnaires, staff will receive information regarding the study and that participation is voluntary. The questionnaires will be distributed in hand and returned in pre-paid envelopes. Two reminders will be sent out to the participants. The project is approved by The Regional Ethical Review Board in Gothenburg, approval number; 355-17. The social Services authorities and the managers from each home agreed to the project. The carers have given their informed consent to attend the study. A project group is established with representatives from the Social Services authorities and the researchers. The implementation of the intervention will be discussed in the project group every second month throughout the study period.

Instruments: This study is planned into three phases. Baseline measures using the Checklist of Challenging Behaviour (CCB). This instrument is translated from English to Swedish and re-translated by experts in the field. It describes 32 observed behaviours relating to CB, for example, verbal, and physical aggression. Scores for items on the instrument range from 1 (the behaviour has not occurred) to 5 (the behaviour occurs daily or more often). The CCB has an acceptable level of content validity and reliability. In the second phase, the intervention will be implemented. The third phase will take place after the intervention with a follow-up period directly after the intervention and after approximately three months in order to analyse effects of the intervention.

At baseline and at follow-up, the instruments will be handed out to the carers to answer. The Job Demand-Control and Social Support (JDC-S) instrument. The JDC-S is a commonly used for investigating psychosocial working environments. This instrument has three major dimensions. First, it measures job demands, which includes psychological stressors such as time pressure, and item scores range from 1 to 4, with higher values indicating higher demands. Second, it measures job control on a scale of 1 to 4, with higher values indicating more perceived control over the job situation. Third, it measures social support, again on a scale of 1 to 4, with higher values indicating higher perceived support from co-workers and managers. In the JDC-S, high demands and low control indicate a high job strain. According to Cronbach's alpha a level of 0.73 for the dimension job demands, 0.52 for job control, and 0.81 for social support was reported.

The Controllability Beliefs Scale (CBS) is a 15-item instrument measuring the attribution of control in situations with CB. This instrument was used to measure carers' values and approaches to people with LD. Items were scored on a 5-point scale with anchored ratings from strongly agree (1) to strongly disagree (5). A two-factor structure, suggesting positive and negative attributions of control, and good internal reliability (Cronbach's alpha for total score = 0.89, 0.92 for the negative subscale and 0.73 for the positive subscale).

The Ways of Coping Questionnaire (WOCQ) measured the use of coping strategies employed by the carers. The instrument was used in this study to measure the intervention's effects in reducing feelings such as shame and guilt in the carers and in strengthening professional care. In this 40-item version of the WOCQ, translated into Swedish, participants were asked to reflect upon how they would manage specific challenging situations. The items were divided into emotion-focused coping skills and problem-focused coping skills. Each subscale was answered on a 4-point Likert scale ranging from (0) does not apply to (3) used a great deal. The instrument was used and tested in a Swedish context with a Cronbach's alpha ranging from 0.63 to 0.89 and has shown acceptable values (> 0.7) on all subscales except for the subscales confrontational coping (0.59) and self-controlling (0.47).

Statistical analysis: Data processing and statistical calculations will be performed in the Statistical Package for Social Sciences (SPSS 23) statistics. Proportions will be compared to the chi-square test. The mean values between the groups will be compared by t-test or Mann-Whitney's U-test, as appropriate. Changes in the mean between and in the groups will be compared with paired t-test. Double-sided significance test will be used throughout. Data will be presented at a group level.

ELIGIBILITY:
Inclusion Criteria:

* staff working at special accommodation for people with intellectual disabilities.
* Language: swedish

Exclusion Criteria:

* staff working short-term temporary agencies at the accommodation for people with intellectual disabilities.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in communication- and interactivity skills and ability to handle challenging behaviour after web-based training program | Before intervention, at intervention completion an average of 12 weeks, and for a 3 month follow up after completed intervention.
  Changes in communication- and interactivity skills and ability to handle challenging behaviour after web-based training program with The checklist of Challenging Behaviour

SECONDARY OUTCOMES:
Ways of Coping Questionnaire | Before intervention, at intervention completion an average of 12 weeks, and for a 3 month follow up after completed intervention.
  Change in coping strategies and practical problem solving with Ways of Coping Questionnaire (WOCQ). Measuring use of coping strategies employed by the carers. The instrument was used in this study to measure the intervention's effects in reducing feelings such as shame and guilt in the carers and in strengthening professional care. In this 40-item version participants were asked to reflect upon how they would manage specific challenging situations. The items were divided into emotion-focused coping skills and problem-focused coping skills. Each subscale was answered on a 4-point Likert scale ranging from (0) does not apply to (3) used a great deal.
The Job Demand-Control and Social Support | Before intervention, at intervention completion an average of 12 weeks, and for a 3 month follow up after completed intervention.
  The Job Demand-Control and Social Support (JDC-S). The instrument has three major dimensions. First, it measures job demands, which includes psychological stressors such as time pressure, and item scores range from 1 to 4, with higher values indicating higher demands. Second, it measures job control on a scale of 1 to 4, with higher values indicating more perceived control over the job situation. Third, it measures social support, again on a scale of 1 to 4, with higher values indicating higher perceived support from co-workers and managers. In the JDC-S, high demands and low control indicate a high job strain.
The Controllability Belief Scale | Before intervention, at intervention completion an average of 12 weeks, and for a 3 month follow up after completed intervention.
  Changes in values and approaches to reduce challenging behavior with The Controllability Belief Scale. The Controllability Beliefs Scale (CBS) is a 15-item instrument measuring the attribution of control in situations with CB. This instrument was used to measure carers' values and approaches to people with LD. Items were scored on a 5-point scale with anchored ratings from strongly agree (1) to strongly disagree (5). A two-factor structure, suggesting positive and negative attributions of control, and good internal reliability (Cronbach's alpha for total score = 0.89, 0.92 for the negative subscale and 0.73 for the positive subscale).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Antonsson, Phd, Principal Investigator — Umea University; Catrin Alverbratt, Phd, Principal Investigator — University West
Locations (1):
- University West, Trollhättan, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonsson H, Graneheim UH, Isaksson U, Astrom S, Lundstrom MO. Evaluation of a Web-Based Training Program for Professional Carers Working With People With Learning Disabilities and Challenging Behavior: A Pilot Study with SSED-Design. Issues Ment Health Nurs. 2016 Oct;37(10):734-743. doi: 10.1080/01612840.2016.1189636. Epub 2016 Jun 28. PMID 27351080
- [Background] Farrell GA, Shafiei T, Salmon P. Facing up to 'challenging behaviour': a model for training in staff-client interaction. J Adv Nurs. 2010 Jul;66(7):1644-55. doi: 10.1111/j.1365-2648.2010.05340.x. Epub 2010 May 21. PMID 20497267
- [Background] Farrell GA, Salmon P. Challenging behaviour: an action plan for education and training. Contemp Nurse. 2009 Dec-2010 Jan;34(1):110-8. doi: 10.5172/conu.2009.34.1.110. PMID 20230177
- [Background] Jenkins R, Rose J, Jones T. The Checklist of Challenging Behaviour and its relationship with the Psychopathology Inventory for Mentally Retarded Adults. J Intellect Disabil Res. 1998 Aug;42 ( Pt 4):273-8. doi: 10.1046/j.1365-2788.1998.00131.x. PMID 9786441
- [Background] Joyce T, Ditchfield H, Harris P. Challenging behaviour in community services. J Intellect Disabil Res. 2001 Apr;45(Pt 2):130-8. doi: 10.1046/j.1365-2788.2001.00331.x. PMID 11298252
- [Background] Sanne B, Mykletun A, Dahl AA, Moen BE, Tell GS. Testing the Job Demand-Control-Support model with anxiety and depression as outcomes: the Hordaland Health Study. Occup Med (Lond). 2005 Sep;55(6):463-73. doi: 10.1093/occmed/kqi071. Epub 2005 Apr 21. PMID 15845554
- [Background] Pellfolk TJ, Gustafson Y, Bucht G, Karlsson S. Effects of a restraint minimization program on staff knowledge, attitudes, and practice: a cluster randomized trial. J Am Geriatr Soc. 2010 Jan;58(1):62-9. doi: 10.1111/j.1532-5415.2009.02629.x. PMID 20122041
- [Background] Dagnan D, Hull A, McDonnell A. The controllability beliefs scale used with carers of people with intellectual disabilities: psychometric properties. J Intellect Disabil Res. 2013 May;57(5):422-8. doi: 10.1111/j.1365-2788.2012.01554.x. Epub 2012 Apr 4. PMID 22471440
- [Background] Folkman S, Moskowitz JT. Coping: pitfalls and promise. Annu Rev Psychol. 2004;55:745-74. doi: 10.1146/annurev.psych.55.090902.141456. PMID 14744233
- [Background] Folkman S, Lazarus RS. The relationship between coping and emotion: implications for theory and research. Soc Sci Med. 1988;26(3):309-17. doi: 10.1016/0277-9536(88)90395-4. PMID 3279520
- [Background] Padyab, Backteman-Erlanson & Brulin. Burnout, Coping, Stress of Conscience and Psychosocial Work Environment among Patrolling Police Officers Journal of Police and Criminal Psychology December 2016, Volume 31, Issue 4, pp 229-237|
- [Background] Dagnan, D., Grant, F., & McDonnell, A. (2004). Understanding challenging behaviour in older people; the development of the Controllability Beliefs Scale. Behavioural and Cognitive Psychotherapy, 32, 501-506.
- [Background] Gore, N., & Umizawa, H. (2011). Challenging behavior training for teaching staff and family carers of children with intellectual disabilities: A preliminary evaluation. Journal of Policy and Practice in Intellectual Disabilities, 8, 266-275.
- [Background] Harris, P., Humphreys, J., & Thomson, G. (1994). A checklist of challenging behaviour: The development of a survey instrument. Mental Handicap Research, 7, 118-133
- [Background] Karasek, R., & Theorell, T. (1992). Healthy work: Stress, productivity and the reconstruction of working life. New York, NY: Basic Books.
- [Background] Mills S, Rose J. The relationship between challenging behaviour, burnout and cognitive variables in staff working with people who have intellectual disabilities. J Intellect Disabil Res. 2011 Sep;55(9):844-57. doi: 10.1111/j.1365-2788.2011.01438.x. Epub 2011 Jul 5. PMID 21726318
- [Derived] Truong AT, Winman T, Ekstrom-Bergstrom A. Studying intraprofessional and interprofessional learning processes initiated by an educational intervention applying a qualitative design with multimethod approach: a study protocol. BMJ Open. 2022 Apr 18;12(4):e058779. doi: 10.1136/bmjopen-2021-058779. PMID 35437255